CLINICAL TRIAL: NCT06814223
Title: Preventive Antibiotic Treatment Before Insertion or Exchange of Tunneled Cuffed Catheters in Hemodialysis Patients to Prevent Early Catheter-Related Infections
Brief Title: Using Antibiotics to Prevent Infections in Hemodialysis Patients During Catheter Placement
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Etty Kruzel-Davila, Director of the Nephrology Department, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0122-24- NHR
Record Dates: First submitted 2025-01-26; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infection Catheter-Related
MeSH Terms: conditions — Catheter-Related Infections | interventions — Cefazolin; Gentamicins

STUDY DESIGN:
Intervention Model Description: This prospective, randomized study will include patients from the hemodialysis unit at the Galilee Medical Center and community-based hemodialysis units. Eligible patients will have one or more of the following high-risk factors: femoral tunneled catheter placement, atrial fibrillation, and/or heart failure. Patients will be hospitalized for the insertion of a new tunneled catheter or the replacement of an existing malfunctioning tunneled catheter.
  Patients with an elevated risk of infection will be randomly assigned to two groups using stratification for new catheter placement versus catheter replacement. Fifty percent of the high-risk patients will receive prophylactic antibiotics targeting gram-positive and gram-negative bacteria 1 hour prior catheter insertion. The antibiotic regimen will include:
  • Cefamezine / vancomycin (2 grams)and gentamicin (80 mg) administered intravenously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PROPHYLACTIC ANTIBIOTIC (Active Comparator): Patients with an elevated risk of infection will be randomly assigned to two groups using stratification for new catheter placement versus catheter replacement. Fifty percent of the high-risk patients will receive prophylactic antibiotics targeting gram-positive and gram-negative bacteria. The antibiotic regimen will include:
  * Cefamezine (2 grams) and gentamicin (80 mg) administered intravenously.
  * Patients with penicillin allergies, a history of methicillin-resistant Staphylococcus aureus (MRSA) infection, or known MRSA colonization will receive vancomycin (2 grams).
  Interventions: Drug: • Cefamezine (2 grams) and gentamicin (80 mg) administered intravenously. • Patients with penicillin allergies, a history of methicillin-resistant Staphylococcus aureus (MRSA) infection, or known MRSA
- No (No Intervention): No prophylactic antibiotic before catheter insertion

INTERVENTIONS:
Drug: • Cefamezine (2 grams) and gentamicin (80 mg) administered intravenously. • Patients with penicillin allergies, a history of methicillin-resistant Staphylococcus aureus (MRSA) infection, or known MRSA — Patients with an elevated risk of infection will be randomly assigned to two groups using stratification for new catheter placement versus catheter replacement. Fifty percent of the high-risk patients will receive prophylactic antibiotics targeting gram-positive and gram-negative bacteria. The antibiotic regimen will include:
  * Cefamezine (2 grams) and gentamicin (80 mg) administered intravenously.
  * Patients with penicillin allergies, a history of methicillin-resistant Staphylococcus aureus (MRSA) infection, or known MRSA colonization will receive vancomycin (2 grams).
  Arms: PROPHYLACTIC ANTIBIOTIC

SUMMARY:
The goal of this clinical trial is to determine if prophylactic antibiotic treatment can reduce the incidence of early catheter-related infections in hemodialysis patients at high risk, including those with femoral catheter placement, atrial fibrillation, or heart failure.

The main questions it aims to answer are:

1. Will prophylactic antibiotic administration reduce catheter-related infections by 50% within 45 days of catheter insertion?
2. Will this intervention decrease the rate of secondary complications such as metastatic infections, cardiovascular morbidity, and mortality?

Researchers will compare patients receiving prophylactic antibiotics (e.g., cefamezine and gentamicin, or vancomycin for high-risk individuals) to those not receiving antibiotics, to assess the difference in infection rates and associated complications.

Participants :

* Be randomized into two groups: one receiving prophylactic antibiotics and one without antibiotics before catheter placement or replacement.
* Undergo follow-up for 45 days to monitor for catheter-related infections and secondary complications.

This study will provide critical data to evaluate whether targeted prophylactic antibiotic treatment should become standard practice for high-risk hemodialysis patients.

DETAILED DESCRIPTION:
Hemodialysis patients undergo renal replacement therapy using vascular access, with an arteriovenous fistula being the ideal access. However, a significant proportion of patients initiate hemodialysis using tunneled catheters, with a gradual decline in catheter use over the following months. According to the United States Renal Data System (USRDS), 74% of patients begin hemodialysis using a catheter, and approximately 20% still use a catheter one year after starting dialysis. Data from dialysis units in France, reported by the Renal Epidemiology and Information Network (REIN), indicate that 56% of patients start hemodialysis using a tunneled catheter.1,2 Catheter-related infections are common complications among chronic hemodialysis patients, contributing to increased morbidity, hospitalizations, and mortality.3,4 Infection is the second most common cause of death among patients with end-stage renal disease, and the use of central venous catheters is associated with increased all-cause and infection-specific mortality.5 According to a study conducted in U.S. dialysis units, the infection rate for tunneled catheters was 8.4 per 100 patient-months. Catheter-related infections can have severe consequences, including prolonged and recurrent hospitalizations, ICU admissions, and metastatic infections such as endocarditis, osteomyelitis, spinal abscesses, and septic arthritis.7,8 Numerous risk factors for catheter-related infections have been identified. A retrospective study examining risk factors for catheter-related infections in 130 patients identified factors such as methicillin-resistant Staphylococcus aureus (MRSA) carriage, bacteremia, or bacteriuria within three months prior to catheter insertion.9 Additional risk factors identified in a meta-analysis of hospitalized patients, including ICU settings, included advanced age, diabetes, a history of catheter-related infections, hypertension, dialysis duration, catheter vein location, catheter indwelling time, multiple catheter insertions, CD4+ T-cell count, albumin level, C-reactive protein (CRP), hemoglobin level, procalcitonin level, and APACHE II scores.10 Moreover, infections have been clearly linked to an increased risk of cardiovascular events, with significant implications for morbidity and mortality in hemodialysis patients, who are already at high risk for both.11,12 Based on the authors clinical observations in the hemodialysis unit at the Galilee Medical Center, the authors identified patients who developed early catheter-related infections (within 45 days of catheter insertion).

A retrospective analysis was conducted on 204 hemodialysis patients who underwent tunneled catheter placement at the Galilee Medical Center between 2020 and 2022. Early catheter-related infections, defined as infections occurring within 45 days of catheter insertion, were documented in 20% (n = 41) of patients.

Multivariate analysis identified the following significant independent risk factors for early tunneled catheter-related infections: Femoral catheter placement: Odds Ratio (OR) = 8.2, p = 0.022, Chronic atrial fibrillation: OR = 8.2, p = 0.022 and Heart failure: OR = 4.9, p = 0.013. The findings suggest a potential benefit of targeted prophylactic antibiotic administration for high-risk patients identified in this study, including those with femoral catheters, atrial fibrillation, and heart failure.

Supporting our findings, an analysis of approximately six million patients hospitalized for sepsis in the U.S. demonstrated that patients with atrial fibrillation had worse prognoses, including prolonged hospital stays, higher treatment costs, and increased all-cause mortality.13 Early catheter-related infection is defined as an infection occurring within 45 days of catheter insertion.14,15 No studies have been published specifically addressing risk factors for early tunneled catheter-related infections. Furthermore, according to the National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines, there is no recommendation for prophylactic antibiotic administration prior to tunneled catheter insertion in dialysis patients.16 Based on these findings, the authors decided to conduct a pragmatic study in our hemodialysis unit to evaluate whether administering prophylactic antibiotics to patients with identified risk factors (femoral catheter placement, atrial fibrillation, and heart failure) can reduce the occurrence of early tunneled catheter-related infections.

Research Rationale Acute infectious diseases are a common complication among hemodialysis patients. Invasive procedures, such as the insertion or replacement of tunneled catheters, significantly increase the risk of early catheter-related infections. Infectious diseases in this population often lead to hospitalizations and can result in severe cardiovascular complications and even mortality.

Given the lack of formal guidelines recommending prophylactic antibiotic administration for hemodialysis patients prior to tunneled catheter insertion, and based on clear findings of risk factors for developing this complication, the authors aim to investigate whether prophylactic antibiotic administration can reduce the likelihood of developing catheter-related infections after catheter insertion.

the authors hypothesize that previous studies did not provide prophylactic antibiotics to defined high-risk groups, and therefore, administering prophylactic antibiotics to a defined high-risk population, as identified in the authors' earlier research, could reduce the incidence of early bloodstream infections following tunneled catheter insertion.

If prophylactic antibiotic administration is found to reduce this complication, it will prompt a change in the antibiotic policy for high-risk patients undergoing tunneled catheter insertion in the hemodialysis unit at the Galilee Medical Center. These findings would also be reported in the global scientific literature.

Study Objectives The study will be a prospective, randomized trial with participants assigned randomly using computer-generated allocation. Prophylactic antibiotic treatment will be administered to 50% of patients identified as high-risk based on the following criteria: femoral catheter placement, atrial fibrillation, and/or heart failure.

Research Hypothesis:

Prophylactic antibiotic administration will reduce the incidence of catheter-related infections by 50% following tunneled catheter insertion.

Research Methodology This prospective, randomized study will include patients from the hemodialysis unit at the Galilee Medical Center and community-based hemodialysis units. Eligible patients will have one or more of the following high-risk factors: femoral tunneled catheter placement, atrial fibrillation, and/or heart failure. Patients will be hospitalized for the insertion of a new tunneled catheter or the replacement of an existing malfunctioning tunneled catheter.

Patients with an elevated risk of infection will be randomly assigned to two groups using stratification for jugular/subclavian catheter insertions versus femoral catheter insertion. Fifty percent of the high-risk patients will receive prophylactic antibiotics targeting gram-positive and gram-negative bacteria. The antibiotic regimen will include:

* Cefamezine (2 grams) and gentamicin (80 mg) administered intravenously 1 hour before the procedure.
* Patients with penicillin allergies, a history of methicillin-resistant Staphylococcus aureus (MRSA) infection, or known MRSA colonization will receive vancomycin (2 grams) instead of Cefamezine.

Primary Endpoint • Early catheter-related infection, defined as an infection occurring within 45 days of tunneled catheter insertion.

Secondary Endpoints

* Metastatic infection complications, including endocarditis and osteomyelitis.
* Cardiovascular morbidity (MACE-major adverse cardiac events) within 90 days after catheter insertion: Acute myocardial infarction, stroke, heart failure and cardiovascular death Research Hypothesis Prophylactic antibiotic administration will reduce the incidence of catheter-related infections by 50% following tunneled catheter insertion.

Study Participants Population

The study will include hemodialysis patients with one or more of the following conditions:

* Heart failure
* Atrial fibrillation
* Use of a femoral tunneled catheter requiring replacement or the insertion of a new tunneled catheter for hemodialysis.

Demographics

* Age range: ≥ 18 years
* Gender: Male and female Inclusion Criteria
* Hemodialysis patients diagnosed with atrial fibrillation and/or heart failure and/or using a femoral tunneled catheter.
* Patients scheduled for new tunneled catheter placement or replacement of an existing tunneled catheter.
* Patients who have signed informed consent to participate in the study. Exclusion Criteria
* Hemodialysis patients unable to provide informed consent and requiring a legal guardian.
* Patients undergoing prolonged antibiotic therapy prior to tunneled catheter insertion.

Withdrawal Criteria

• None specified (not applicable).

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients scheduled for new tunneled catheter placement or replacement of an existing tunneled catheter.
* Prior diagnosis of at least one of the following conditions:

  1. Atrial fibrillation
  2. Heart failure
  3. Femoral tunneled catheter

     * Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

* • Hemodialysis patients unable to provide informed consent and requiring a legal guardian.

  * Patients undergoing prolonged antibiotic therapy prior to tunneled catheter insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Early catheter-related infection, defined as an infection occurring within 45 days of tunneled catheter insertion. | 45 days after chatter insertion
  • Early catheter-related infection, defined as an infection occurring within 45 days of tunneled catheter insertion. (present/absent): These data will be collected from the patient's medical record based on clinical documentation of infection, including positive blood cultures.

SECONDARY OUTCOMES:
Metastatic infection | 90 days after catheter infection
  •Metastatic infection: endocarditis, endovascular infection and osteomyelitis. Present/absent: These data will be collected from the patient's medical record based on clinical documentation of these complications.
Major adverse cardiovascular events (MACE): | 90 days after catheter insertion
  Acute myocardial infarction (AMI), stroke, heart failure and cardiovascular death (yes/no) These data will be collected from the patient's medical record based on clinical documentation of these complications..
Mortality | 90 days after catheter insertion.
  All cause mortality- yes/no. This endpoint will be collected from the patient's medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Center, Nahariya, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
All anonymized data collected during the study will be made available upon reasonable request. This ensures transparency and allows for independent validation of the findings while protecting participant privacy. Identifiable information will be removed, and data will only be shared in a de-identified format, ensuring that participants cannot be traced back based on the shared data. Access to the anonymized dataset will require approval from the principal investigator to ensure appropriate use and adherence to ethical standards.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] 1. https://usrds-adr.niddk.nih.gov/2023/end-stage-renal-disease/4-vascular-access, 2021 2. Lassalle M, Monnet E, Ayav C, Hogan J, Moranne O, Couchoud C, et al. 2017 annual report digest of the renal epidemiology information network (REIN) registry. Transpl. Int. 2019;32(9):892-902. doi: 10.1111/tri.13466. 3. Arhuidese IJ, Cooper MA, Rizwan M, Nejim B, Malas MB. Vascular access for hemodialysis in the elderly. J. Vasc. Surg. 2019;69(2):517-525. doi: 10.1016/j.jvs.2018.05.219. 4. Ravani P, Palmer SC, Oliver MJ, Quinn RR, MacRae JM, Tai DJ, et al. Associations between hemodialysis access type and clinical outcomes: A systematic review. J. Am. Soc. Nephrol. 2013;24(3):465-473. doi: 10.1681/ASN.2012070643. 5. Aslam S, Vaida F, Ritter M, Ravindra L. Systematic review and meta-analysis on management of hemodialysis catheter-related bacteremia. J. Am. Soc. Nephrol. 2014;25(12):2927-2941. doi: 10.1681/ASN.2013091009. 6. Tokars JI, Miller ER, Stein G. New national surveillance system for hemodialysis associated infections: initial results. Am J Infect Control. 2002;30(5):288-295. 7. Chavers BM, Solid CA, Gilbertson DT, Collins AJ. Infection-related hospitalization rates in pediatric versus adult patients with end-stage renal disease in the United States. J Am Soc Nephrol. 2007 Mar;18(3):952-9. 8. Farrington CA, Allon M. Complications of Hemodialysis Catheter Bloodstream Infections: Impact of Infecting Organism. Am J Nephrol. 2019;50(2):126-132. 9. Delistefani, F., Wallbach, M., Müller, G.A. et al. Risk factors for catheter-related infections in patients receiving permanent dialysis catheter. BMC Nephrol 20, 199 (2019). 10. Huajie Guo , Ling Zhang ,Hua He , Lili Wang. Risk factors for catheter-associated bloodstream infection in hemodialysis patients: A meta-analysis. Published: March 27, 2024. Crossref DOI link: https://doi.org/10.1371/journal.pone.0299715 11. Pyry N. Sipilä, Joni V. Lindbohm, G. David Batty, Nelli Heikkilä, Jussi Vahtera, Sakari Suominen, Ari Väänänen
- Available data/document: Study Protocol — https://my.health.gov.il/CliniTrials/Pages/Home.aspx